CLINICAL TRIAL: NCT01840917
Title: Heart Rate Variability in the Course of Acute Uncomplicated Diverticulitis
Brief Title: Heart Rate Variability During Acute Diverticulitis
Status: Completed | Type: Observational
Sponsor: Herlev Hospital (Other)
Collaborators: Lundbeck Foundation (Other)
Responsible Party: Principal Investigator, Ismail Gögenür, Senior resident and D.Sc., Herlev Hospital
Other Study IDs: CHU-4
Record Dates: First submitted 2013-04-13; First posted 2013-04-26 (Estimated); Last update posted 2014-02-25 (Estimated); Status verified 2014-02

CONDITIONS: Acute Diverticulitis

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- acute uncomplicated diverticulitis: CT-verified acute uncomplicated diverticulitis managed by antibiotics

SUMMARY:
The purpose of this study is to investigate heart rate variability during Acute uncomplicated diverticulitis by ECG-monitor (Holter), the investigators hypothesis is the inflammation causes a decrease of High Frequency(HF)-power component of heart rate variability and this correlates with sleep quality and daytime fatigue.

DETAILED DESCRIPTION:
An increasing number of studies have shown that circadian variation in the excretion of hormones, the sleep-wake cycle, the core body temperature, the tone of the autonomic nervous system and the activity rhythm are important both in health and disease processes. The investigators are interested in investigating the heart rate variability (HRV) during an acute surgical non-inflammatory condition, and to exam whether there are correlations between: HRV and sleep stages, HRV and cytokine levels in blood and HRV and subjective fatigue.

Following methods will be applied

Device: Holter monitor - Medilog AR12 (Oxford Instruments, Oxford, England)

Other: Karolinska Sleepiness Scale

Other: Physical Fatigue Scale

Device: Polysomnograph - Embla Titanium (Natus Medical Incorporated, USA)

Procedure: Plasma cytokines (IL-2, IL-6 and TNF(tumor necrosis factor)-alfa)

Procedure: Plasma CRP(C reactive protein) and leukocytes

ELIGIBILITY:
Inclusion Criteria:

* CT-verified diverticulitis patients managed by antibiotic treatment at Herlev Hospital
* Pain and fever occurred less than 72 hours prior to the admission
* ASA (American Society of Anesthesiologists) score I to III

Exclusion Criteria:

* Surgical intervention needed
* Complicated diverticulitis
* Complications in relation to diverticulitis
* Pain and fever occurred more than 72 hours prior to the admission
* In anticoagulant treatment and heart rate control treatment
* Known Autoimmune disease
* Known medically treated sleep-disorder (insomnia, restless legs etc.) and sleep apnea
* Shift-work or jetlag
* Daily use of opioid, psychopharmaca, opioids or anxiolytics (including Hypnotics)
* Known psychiatry conditions in treatment with psychopharmaca
* Daily alcohol intake of more than 5 units or drug abuse
* Missing written consent
* Diabetes Mellitus
* Predicted bad compliance
* Pregnant or breast-feeding
* Urine or fecal incontinence
* Severe kidney disease
* Current cancer

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 16 x Acute uncomplicated diverticulitis (Hansen and stock stage 1) patients aged 18-75 years managed by antibiotic treatment at Herlev Hospital
Sampling Method: Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2013-04; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Heart-rate variability changes during the acute uncomplicated diverticulitis compared to the baseline levels at 30th night where the condition has been cured | 1st, 2nd and 30th night following the admission
  Heart-rate variability measured by Holter monitor and a following analysis of frequency and time domain parameters.

SECONDARY OUTCOMES:
changes in plasma cytokine levels during the acute uncomplicated diverticulitis from the baseline levels at 30th day (remission) | 1st, 2nd and 30th days following the admission
  the blood sample is taken at night before sleep time. the cytokines are measured with ELISA-kit
change in Sleep data during the acute diverticulitis from baseline Sleep data at remission (30th day) | 1st, 2nd and 30th days following the admission
  Sleep data is measured by Polysomnography and sleep is categorized into sleep stages (awake, stage 1, 2, REM-sleep and SWS-sleep)

CONTACTS AND LOCATIONS:
Overall Officials: Ismail Gögenur, M.D., Principal Investigator — University of Copenhagen, Herlev Hospital
Locations (1):
- Department D, Herlev Hospital, Herlev, Copenhagen, Denmark